CLINICAL TRIAL: NCT00117949
Title: An Open-Label, Multi-Center, Ascending, Single Dose Study Investigating the Pharmacokinetics, Pharmacodynamics and Safety of FE200486
Brief Title: Study Investigating the Pharmacokinetics, Pharmacodynamics and Safety of FE200486
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Clinical Development Support, Ferring Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS06
Record Dates: First submitted 2005-06-30; First posted 2005-07-11 (Estimated); Results first posted 2009-06-05 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen ablation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Degarelix 40 mg (Experimental): Degarelix 40 mg (10 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 80 mg (Experimental): Degarelix 80 mg (20 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 120 mg (Experimental): Degarelix 120 mg (30 mg/mL)
  Interventions: Drug: Degarelix
- Degarelix 160 mg (Experimental): Degarelix 160 mg (40 mg/mL)
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — One dose (2 x 2 mL) of degarelix 40 mg (10 mg/mL), subcutaneous injection.
  Other Names: FE200486
  Arms: Degarelix 40 mg
Drug: Degarelix — One dose (2 x 2 mL) of degarelix 80 mg (20 mg/mL), subcutaneous injection.
  Other Names: FE200486
  Arms: Degarelix 80 mg
Drug: Degarelix — One dose (2 x 2 mL) of degarelix 120 mg (30 mg/mL), subcutaneous injection.
  Other Names: FE200486
  Arms: Degarelix 120 mg
Drug: Degarelix — One dose (2 x 2 mL) of degarelix 160 mg (40 mg/mL), subcutaneous injection.
  Other Names: FE200486
  Arms: Degarelix 160 mg

SUMMARY:
Population pharmacokinetic and pharmacodynamic data from Study FE200486 CS06 and FE200486 CS02 provided further knowledge of the optimal dose regimens for FE200486 (degarelix). Both studies were to guide dose selection for phase III. In addition, safety and tolerance data were generated.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following inclusion criteria before entry into the study:

* Has given written consent before any study related activity is performed (A study related activity is defined as any procedure that would not have been performed during the normal management of the patient.)
* Is a male patient with histologically proven adenocarcinoma of the prostate (all stages) in whom endocrine treatment is indicated, except for neoadjuvant hormonal therapy. For patients, prostate-specific antigen (PSA) increases on two consecutive determinations at least 2 weeks apart prior to Visit 1 must be documented.
* Is at least 18 years.
* Has an ECOG score of 2.
* Has a baseline testosterone level within the age specific normal range as measured by the central laboratory.
* Has a PSA value of 2 ng/mL as measured by the central laboratory.
* Has a life expectancy of at least 6 months.

Exclusion Criteria:

Any patient meeting one or more of the following exclusion criteria will not be entered into the study:

* Previous or present hormonal management of prostate cancer (surgical castration or other hormonal manipulation, e.g. GnRH agonists, GnRH antagonists, antiandrogens, estrogens, PC-Spec) except for neoadjuvant hormonal therapy of < 6 months duration and completed > 6 months prior to Visit 1.
* Requires hormonal therapy for neoadjuvant purposes.
* Is recently (within the last 12 weeks preceding Visit 1) or presently treated with any other drug modifying the testosterone level or function.
* Is considered to be a candidate for curative therapy, i.e., radical prostatectomy or radiotherapy within 6 months after Visit 1.
* Has a history of severe asthma requiring daily treatment with inhalation steroids, angioedema or anaphylactic reactions.
* Has hypersensitivity towards any component of the investigational product.
* Has had a cancer disease within the last 10 years except for prostate cancer, and surgically removed basocellular or squamous cell carcinoma of the skin.
* Has a clinically significant neurologic, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, dermatological or infectious disorder or any other condition, including excessive alcohol or drug abuse, which may interfere with trial participation, or which may affect the conclusion of the study, as judged by the investigator.
* Any clinically significant laboratory abnormalities which, in the judgment of the investigator, would interfere with the patient's participation in this study or evaluation of study results (liver transaminases must be within normal limits).
* Has a mental incapacity or language barrier precluding adequate understanding or co-operation.
* Has received an investigational drug within the last 12 weeks preceding Visit 1.
* Has previously participated in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2002-04; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (12):
- United States (12):
  - Advanced Urology Medical Center, Anaheim, California
  - South Orange County Medical Research Center, Laguna Woods, California
  - San Bernardino Urological Associates Medical Group, San Bernardino, California
  - Western Clinical Research, Torrance, California
  - Urology Associate PC', Denver, Colorado
  - SW Florida Urological Associates, Fort Myers, Florida
  - Pinellas Urology, Inc., St. Petersburg, Florida
  - Drs. Werner, Murdock & Francis, PA, Greenbelt, Maryland
  - Nevada Urology Associates, Reno, Nevada
  - Urology Specialists of Oklahoma, Inc., Tulsa, Oklahoma
  - Urology Clinics of NorthTexas, PA, Dallas, Texas
  - Urology San Antonio Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were followed until they met a pre-defined criterion for insufficient testosterone or prostate-specific antigen (PSA).
Period: Overall Study
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Started | 10 (Dose level terminated prematurely due to inadequate testosterone response) | 24 | 24 | 24
Completed | 0 | 0 | 0 | 0
Not Completed | 10 | 24 | 24 | 24
Not completed — Testosterone >1.0 ng/mL | 10 | 18 | 17 | 15
Not completed — Testosterone 0.5 - 1.0 ng/mL | 0 | 1 | 3 | 2
Not completed — Prostate-specific antigen increase >=25% | 0 | 1 | 1 | 2
Not completed — PSA increase >=10ng/mL | 0 | 1 | 1 | 0
Not completed — PSA reduction <=50% | 0 | 2 | 2 | 4
Not completed — Hepatic abnormalities | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg | Total
Number analyzed (Participants) | 10 | 24 | 24 | 24 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2 | 4 | 8
  >=65 years | 9 | 23 | 22 | 20 | 74
Age Continuous [Mean (Standard Deviation); unit: years] | 72.0 (5.7) | 77.5 (6.4) | 75.9 (5.8) | 74.7 (8.4) | 75.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 10 | 24 | 24 | 24 | 82
Race/Ethnicity, Customized [Number; unit: participants]
  Oriental/Asian | 0 | 0 | 0 | 0 | 0
  Black | 2 | 1 | 2 | 1 | 6
  Caucasian | 5 | 23 | 15 | 20 | 63
  Other | 3 | 0 | 7 | 3 | 13
Gleason score [Number; unit: participants] — The Gleason score is a system of grading the aggressiveness of the prostate cancer and how fast it is likely to grow and spread. Scale is 2-10, with low numbers being the least aggressive and 10 being the most aggressive.
  participants
    Unknown | 0 | 1 | 0 | 0 | 1
    2-4 | 1 | 1 | 1 | 0 | 3
    5-6 | 3 | 14 | 12 | 13 | 42
    7-10 | 6 | 8 | 11 | 11 | 36
Stage of prostate cancer [Number; unit: participants] — Prostate cancer stage was classified to describe the extent of cancer. Localized refers to tumors without involvement of lymph nodes or metastasis. Advanced localized can be larger tumors that may involve the lymph nodes but no metastasis. Metastatic are more advanced cancers that are spreading beyond the original tumor.
  participants
    Localized | 5 | 11 | 12 | 10 | 38
    Locally advanced | 0 | 6 | 5 | 5 | 16
    Metastatic | 2 | 4 | 2 | 2 | 10
    Not classifiable | 3 | 3 | 5 | 7 | 18
Body mass index [Mean (Standard Deviation); unit: kilogram per square meter] — Body mass index is a measure of body fat based on height and weight.
  kilogram per square meter | 26.70 (5.72) | 26.61 (3.55) | 27.22 (3.16) | 26.64 (3.38) | 26.70 (5.72)
Serum prostate-specific antigen levels [Median (Full Range); unit: nanogram per milliliter] | 9.30 [2.3 to 36.3] | 13.40 [3.6 to 765] | 9.10 [2.2 to 50.9] | 6.40 [2.2 to 154] | 9.35 [2.2 to 765]
Serum testosterone levels [Median (Full Range); unit: nanogram per milliliter] | 3.98 [2.29 to 5.31] | 4.10 [1.79 to 8.53] | 3.96 [2.02 to 7.22] | 3.89 [1.79 to 8.53] | 3.93 [1.79 to 8.53]
Time since prostate cancer diagnosis [Mean (Standard Deviation); unit: days] — The mean number of days since a diagnosis of prostate cancer was made for the patients in each study group.
  days | 851 (1077) | 954 (1328) | 1609 (1836) | 1095 (1385) | 1181 (1494)
Weight [Mean (Standard Deviation); unit: kilogram] | 78.97 (11.73) | 81.73 (11.50) | 80.77 (12.83) | 81.40 (14.36) | 81.01 (12.61)

OUTCOME MEASURES:

1. Primary Outcome: Time to Meet Insufficient Testosterone Response
Description: Figures in the table are Kaplan-Meier estimates of the time to meeting insufficient testosterone response. Insufficient testosterone response was defined as testosterone >1.0 ng/mL at one visit or testosterone 0.5-1.0 at two consecutive visits.
Time Frame: 3 months
Population: Patients who withdrew without meeting the insufficient testosterone (T) suppression criteria were censored as of the time for last available T measurement prior to discontinuation. For the 40 mg group the 95% confidence interval around the time estimate was non-estimable and no statistical analysis is presented (the estimate was 14 days).
Measure: Median (Full Range); unit: days
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Number analyzed (Participants) | 10 | 24 | 24 | 24
days | 14 [14 to 70] | 77 [14 to 140] | 98 [14 to 219] | 28 [14 to 126]
Statistical Analysis 1: Comparison: Degarelix 40 mg vs Degarelix 80 mg vs Degarelix 120 mg vs Degarelix 160 mg; Test type: Superiority or Other; p < 0.001, Log Rank
Statistical Analysis 2: Comparison: Degarelix 80 mg; Kaplan-Meier estimates of the time to meet insufficient testosterone (T) response; Test type: Superiority or Other; Median days to insufficient T response = 84, 95% CI [35 to 112]
Statistical Analysis 3: Comparison: Degarelix 120 mg; Kaplan-Meier estimates of the time to meet insufficient testosterone (T) response; Test type: Superiority or Other; Median days to insufficient T response = 98, 95% CI [70 to 126]
Statistical Analysis 4: Comparison: Degarelix 160 mg; Kaplan-Meier estimates of the time to meet insufficient testosterone (T) response; Test type: Superiority or Other; Median days to insufficient T response = 35, 95% CI [14 to 98]

2. Secondary Outcome: Time to Testosterone Castration (Testosterone ≤0.5 ng/mL).
Description: Time to testosterone castration was calculated as the number of days from dosing to the first scheduled visit when testosterone was less than 0.5 ng/mL. The figures in the table present the number of participants who were castrated after 1, 3, 7, 14, 21, 28, and 42 days.
Time Frame: 1, 3, 7, 14, 21, 28, 42 days
Population: Half participants in the 40 mg group were not castrated and the median was not calculated (no statistical anaylsis was made). Two participants out of 24 in the 80 mg, 1/24 in the 120 mg, and 3/24 in the 160 mg groups were not castrated. For the 160 mg group the 95% CI was non-estimable and no statistical anaylsis was made.
Measure: Number; unit: days
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Number analyzed (Participants) | 10 | 24 | 24 | 24
days
  1 day | 1 [3 to NA] | 3 [3 to 7] | 11 [1 to 3] | 6 [NA to NA]
  3 days | 3 | 12 | 12 | 14
  7 days | 1 | 2 | 0 | 1
  14 days | 0 | 2 | 0 | 0
  21 days | 0 | 1 | 0 | 0
  28 days | 0 | 1 | 0 | 0
  42 days | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Degarelix 40 mg vs Degarelix 80 mg vs Degarelix 120 mg vs Degarelix 160 mg; Test type: Superiority or Other; p = 0.003, Log Rank; Participants not castrated were censored as of the days from dosing for the last available observation
Statistical Analysis 2: Comparison: Degarelix 80 mg; Kaplan-Meier estimates of the median time to testosterone castration; Test type: Superiority or Other; Median time to castration (days) = 3, 95% CI [3 to 7]
Statistical Analysis 3: Comparison: Degarelix 120 mg; Kaplan-Meier estimates of the time to testosterone castration; Test type: Superiority or Other; Median time to castration (days) = 3, 95% CI [1 to 3]

3. Secondary Outcome: Number of Participants With Sufficient Testosterone Suppression for at Least 84 Days
Description: Sufficient testosterone suppression was defined as not meeting an insufficient testosterone response criterion. Insufficient testosterone response was defined as testosterone >1.0 ng/mL at one visit or testosterone 0.5-1.0 at two consecutive visits.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Number analyzed (Participants) | 10 | 24 | 24 | 24
participants | 0 [0 to 0] | 9 [22.0 to 63.4] | 14 [41.8 to 81.3] | 7 [15.8 to 55.5]
Statistical Analysis 1: Comparison: Degarelix 40 mg; Kaplan-Meier estimates of the percentage of participants with sufficient testosterone suppression; Test type: Superiority or Other; Percentage of participants = 0, 95% CI [0 to 0]
Statistical Analysis 2: Comparison: Degarelix 80 mg; Kaplan-Meier estimates of the percentage of participants with sufficient testosterone suppression; Test type: Superiority or Other; Percentage of participants = 42.7, 95% CI [22 to 63.4]
Statistical Analysis 3: Comparison: Degarelix 120 mg; Kaplan-Meier estimates of the percentage of participants with sufficient testosterone suppression; Test type: Superiority or Other; Percentage of participants = 61.6, 95% CI [41.8 to 81.3]
Statistical Analysis 4: Comparison: Degarelix 160 mg; Kaplan-Meier estimates of the percentage of participants with sufficient testosterone suppression; Test type: Superiority or Other; Percentage of participants = 35.6, 95% CI [15.8 to 55.5]

4. Primary Outcome: Number of Participants With Testostestone Serum Levels Below 0.5 ng/mL for at Least 28 Days
Description: The number of participants suppressed for at least 28 days was defined as the estimated "survival probability" at time=Day 28.
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Number analyzed (Participants) | 10 | 24 | 24 | 24
participants | 1 [0.3 to 44.5] | 17 [48.9 to 87.4] | 19 [57.8 to 92.9] | 13 [32.8 to 74.4]
Statistical Analysis 1: Comparison: Degarelix 40 mg vs Degarelix 80 mg vs Degarelix 120 mg vs Degarelix 160 mg; Test type: Superiority or Other; p = 0.181, Cochran-Armitage Trend Test
Statistical Analysis 2: Comparison: Degarelix 40 mg; Kaplan Meier-estimates of the percentage of participants with testostestone serum levels below 0.5 ng/mL for at least 28 days; Test type: Superiority or Other; Percentage of participants = 10, 95% CI [0.3 to 44.5]
Statistical Analysis 3: Comparison: Degarelix 80 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; Percentage of participants = 70.8, 95% CI [48.9 to 87.4]
Statistical Analysis 4: Comparison: Degarelix 120 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; Percentage of participants = 79.2, 95% CI [57.8 to 92.9]
Statistical Analysis 5: Comparison: Degarelix 160 mg; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; Percentage of participants = 54.2, 95% CI [32.8 to 74.4]

5. Secondary Outcome: Time to 50% Reduction in Prostate-specific Antigen Levels
Description: The time to 50% prostate-specific antigen (PSA) reduction from baseline was defined as the median number of days from dosing to the first visit where a 50% reduction in PSA level was reached.
Time Frame: 3 months
Population: Participants who did not achieve the actual level of reduction were censored as of the time from dosing for the last available observation. In the 40 mg group only two participants reached a 50% reduction in PSA and the Kaplan-Meier estimate could not be calculated (ie no statistical analysis is presented for this group).
Measure: Median (Full Range); unit: days
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Number analyzed (Participants) | 10 | 24 | 24 | 24
days | 10.5 [7 to 14] | 14 [7 to 42] | 14 [7 to 35] | 14 [7 to 42]
Statistical Analysis 1: Comparison: Degarelix 40 mg vs Degarelix 80 mg vs Degarelix 120 mg vs Degarelix 160 mg; Test type: Superiority or Other; p = 0.046, Log Rank
Statistical Analysis 2: Comparison: Degarelix 80 mg; Kaplan-Meier estimates of the time (days) to 50% reduction in PSA; Test type: Superiority or Other; days = 14, 95% CI [14 to 28]
Statistical Analysis 3: Comparison: Degarelix 120 mg; Kaplan-Meier estimates of the time (days) to 50% reduction in PSA; Test type: Superiority or Other; days = 14, 95% CI [14 to 28]
Statistical Analysis 4: Comparison: Degarelix 160 mg; Kaplan-Meier estimates of the time (days) to 50% reduction in PSA; Test type: Superiority or Other; days = 28, 95% CI [14 to 41]

6. Secondary Outcome: Time to 90% Reduction in Prostate-specific Antigen Levels
Description: The time to 90% prostate-specific antigen (PSA) reduction from baseline was defined as the median number of days from dosing to the first visit where a 90% reduction in PSA level was reached.
Time Frame: 3 months
Population: Participants who did not achieve the actual level of reduction were censored as of the time from dosing for the last available observation. In the 40 mg group only one participant reached a 90% reduction in PSA and the Kaplan-Meier estimate could not be calculated (ie no statistical analysis is presented for this group).
Measure: Median (Full Range); unit: days
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Number analyzed (Participants) | 10 | 24 | 24 | 24
days | 28 [28 to 28] | 35 [28 to 98] | 35 [28 to 84] | 31.5 [14 to 56]
Statistical Analysis 1: Comparison: Degarelix 40 mg vs Degarelix 80 mg vs Degarelix 120 mg vs Degarelix 160 mg; Test type: Superiority or Other; p = 0.926, Log Rank
Statistical Analysis 2: Comparison: Degarelix 80 mg; Kaplan-Meier estimates of the time (days) to 90% reduction in PSA; Test type: Superiority or Other; days = 56, 95% CI [35 to 56]
Statistical Analysis 3: Comparison: Degarelix 120 mg; Kaplan-Meier estimates of the time (days) to 90% reduction in PSA; Test type: Superiority or Other; days = 56, 95% CI [35 to 84]
Statistical Analysis 4: Comparison: Degarelix 160 mg; Kaplan-Meier estimates of the time (days) to 90% reduction in PSA; Test type: Superiority or Other; days = 56, 95% CI [35 to 100] — The upper confidence interval limit could not be calculated. For technical reasons it has been entered as 100

7. Secondary Outcome: Liver Function Tests
Description: The number of participants who had abnormal (defined as above upper limit of normal range (ULN)) alanine aminotransferase (ALT) levels, aspartate aminotransferas levels, and bilirubin levels plus the number of participants who had ALT increases >3x ULN and ALT increases >3x ULN with concurrently increased bilirubin >1.5 ULN.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Number analyzed (Participants) | 10 | 24 | 24 | 24
participants
  Abnormal alanine aminotransferase (ALAT) | 0 | 3 | 3 | 6
  Abnormal aspartate aminotransferase | 1 | 11 | 13 | 9
  Abnormal bilirubin | 2 | 0 | 2 | 2
  ALAT >3x upper limit of normal (ULN) | 0 | 1 | 0 | 0
  ALAT >3x ULN, bilirubin >1.5x ULN | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Serious Adverse Events (participants affected / at risk) | 0 | 1 | 1 | 0
Other Adverse Events (participants affected / at risk) | 6 | 18 | 20 | 13
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Small intestinal obstruction (Gastrointestinal disorders) | 0/10 (0) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Chest pain (General disorders) | 0/10 (0) | 1/24 (1) | 0/24 (0) | 0/24 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Degarelix 40 mg | Degarelix 80 mg | Degarelix 120 mg | Degarelix 160 mg
Anaemia (Blood and lymphatic system disorders) | 0/10 (0) | 0/24 (0) | 3/24 (4) | 0/24 (0)
Diabetic retinopathy (Eye disorders) | 1/10 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0)
Diarrhoea (Gastrointestinal disorders) | 0/10 (0) | 1/24 (1) | 2/24 (2) | 0/24 (0)
Constipation (Gastrointestinal disorders) | 0/10 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0)
Haemorrhoids (Gastrointestinal disorders) | 0/10 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0)
Inguinal hernia (Gastrointestinal disorders) | 0/10 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0)
Injection site pain (General disorders) | 0/10 (0) | 2/24 (2) | 3/24 (4) | 1/24 (1)
Fatigue (General disorders) | 1/10 (1) | 2/24 (2) | 0/24 (0) | 2/24 (2)
Injection site pruritus (General disorders) | 0/10 (0) | 2/24 (2) | 1/24 (1) | 0/24 (0)
Chest pain (General disorders) | 0/10 (0) | 2/24 (4) | 0/24 (0) | 0/24 (0)
Nasopharyngitis (Infections and infestations) | 0/10 (0) | 2/24 (2) | 3/24 (3) | 1/24 (1)
Alanine aminotransferase increased (Investigations) | 0/10 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0)
Aspartate aminotransferase increased (Investigations) | 0/10 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0)
Breath sounds abnormal (Investigations) | 1/10 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1/10 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1/10 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0)
Dizziness (Nervous system disorders) | 1/10 (1) | 2/24 (2) | 2/24 (2) | 1/24 (1)
Headache (Nervous system disorders) | 1/10 (1) | 1/24 (1) | 2/24 (2) | 0/24 (0)
Libido decreased (Psychiatric disorders) | 0/10 (0) | 0/24 (0) | 0/24 (0) | 2/24 (2)
Dysuria (Renal and urinary disorders) | 0/10 (0) | 2/24 (2) | 1/24 (1) | 1/24 (1)
Urinary retention (Renal and urinary disorders) | 0/10 (0) | 2/24 (2) | 0/24 (0) | 0/24 (0)
Urine flow decreased (Renal and urinary disorders) | 1/10 (1) | 0/24 (0) | 0/24 (0) | 0/24 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0/10 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0/10 (0) | 2/24 (3) | 0/24 (0) | 0/24 (0)
Hot flush (Vascular disorders) | 2/10 (2) | 12/24 (12) | 5/24 (6) | 5/24 (5)
Hypertension (Vascular disorders) | 0/10 (0) | 0/24 (0) | 2/24 (2) | 0/24 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript.